CLINICAL TRIAL: NCT07190313
Title: Massage: Neuroimaging and Correlates of Response
Brief Title: Massage: Neuroimaging and Correlates of Response - 1-week Study
Acronym: Massage: Neuro
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Mark Rapaport, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB #155218
Record Dates: First submitted 2025-09-08; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: massage, magnetic resonance imaging

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized, single masked study investigating the effects of a single session of Swedish massage therapy (SMT) vs. a light touch (LT) control on brain activity, assessments, and autonomic function in healthy non-psychiatric control subjects.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Of necessity, the coordinator, subjects, and therapists will know their randomized group assignment. Other study staff interacting with participants, including the investigator completing adverse event assessments, will be masked to the treatment assignment. Participants randomized to a treatment arm will be asked not to disclose their assigned treatment to those staff members. The study coordinator and therapists performing the SMT and LT interventions will not discuss subjects' treatment assignment with other staff at any time during the study. The study statistician will perform and report the primary and secondary outcome analyses using masked treatment codes. The non-masked coordinator will have access to the study randomization schedule and may unmask subjects only in the case of emergency, or if necessary, to establish proper follow-up treatment for a condition that arises during the course of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Swedish Massage Therapy (Experimental): The therapist uses non-aromatic cream to facilitate making long strokes over the body. Swedish massage is done with the subject covered by a sheet, a technique called "draping." One part of the body is uncovered, massaged, and then re-draped before moving to another part. The primary techniques used in the research protocol therapy are effleurage, petrissage, kneading, tapotement and thumb friction. These techniques are performed in a very precise, carefully elaborated manner. The session starts with the subject fully draped in a prone position on the massage table and after approximately 22 minutes the subject is instructed to turn to the supine position. Finally, the therapist moves to the head area of the subject, begins working on the shoulders, neck and head using effleurage and thumb friction, and concludes by using light tapotement on the head. The total time for the entire massage is 45 minutes. Subjects randomized to SMT will undergo a single session.
  Interventions: Other: Swedish Massage Therapy
- Light Touch Control (Active Comparator): The Light Touch Control protocol entails the same duration and sequence of procedures as the massage protocol, except that the therapist employs only light-touch hand placement on the subject's body. This condition isolates the effect of the mechanical intervention of SMT. Subjects randomized to LT will undergo a single session.
  Interventions: Other: Light Touch Control

INTERVENTIONS:
Other: Swedish Massage Therapy — The therapist uses non-aromatic cream to facilitate making long strokes over the body. Swedish massage is done with the subject covered by a sheet, a technique called "draping." One part of the body is uncovered, massaged, and then re-draped before moving to another part. The primary techniques used in the research protocol therapy are effleurage, petrissage, kneading, tapotement and thumb friction. These techniques are performed in a very precise, carefully elaborated manner. The session starts with the subject fully draped in a prone position on the massage table and after approximately 22 minutes the subject is instructed to turn to the supine position. Finally, the therapist moves to the head area of the subject, begins working on the shoulders, neck and head using effleurage and thumb friction, and concludes by using light tapotement on the head. The total time for the entire massage is 45 minutes. Subjects randomized to SMT will undergo a single session.
  Arms: Swedish Massage Therapy
Other: Light Touch Control — The Light Touch Control protocol entails the same duration and sequence of procedures as the massage protocol, except that the therapist employs only light-touch hand placement on the subject's body. This condition isolates the effect of the mechanical intervention of SMT. Subjects randomized to LT will undergo a single session.
  Arms: Light Touch Control

SUMMARY:
This study will compare the effects (good or bad) of Swedish massage or light touch therapy on your brain activity, physical responses (like heart rate, blood pressure, breathing rate), and mood and stress. This is a randomized research study. "Randomized" means that participants will be assigned to a study group by chance, like flipping a coin. Participants will be randomized into one of two study groups, and will have an equal chance of being placed in one of the groups: - A single session of Swedish massage therapy - A single session of Light touch therapy At the study visit, the study staff ask about life stressors, medical health, medicine use, and illicit substance use over the past week. The study uses magnetic resonance imaging (MRI) as well as functional MRI (fMRI) to look at the structure and activation of the brain. Participants will undergo two brain scanning sessions, one immediately before and one immediately after the Swedish massage or light touch therapy. The scans will last approximately 45 minutes. During the brain scanning sessions, information on heart rate, blood pressure, temperature and breathing will also be collected.

DETAILED DESCRIPTION:
This is a two-arm, randomized, single masked study investigating the effects of a single session of Swedish massage therapy (SMT) vs. a light touch (LT) control on brain activity, assessments, and autonomic function in non-psychiatric control subjects. The Primary Objective is to identify brain networks activated by SMT vs. LT using resting state fMRI and Functional Connectivity during the neutral/fearful/angry faces task in normal control subjects. The secondary objective is to correlate changes in autonomic measures with resting state fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* aged ≥ 18 and < 65 years old.
* Medically stable
* Psychiatrically healthy as demonstrated by a structured clinical interview that elicits no previous or current Axis I psychopathology
* Ability to lie prone or supine for one hour at a time, given the nature of the massage intervention
* Subjects must have a permanent domicile
* Subjects must be able to comply with the research protocol
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Current (within 3 months of screening visit) nicotine use, illicit drug use, or long-term medication use that, in the opinion of the investigator, could alter the results of the study
* Pregnancy (per participant report, pregnancy testing not done for study)
* Usually is asleep during the daytime (ie due to Working third-shift), or any other behaviors that routinely disrupt normal diurnal (daily) rhythms
* Current (past month) rigorous dieting (defined as <1200 calories per day for ≥2 consecutive days)
* In the month before screening visit, excessive regular use of alcohol, as defined by either of the following, twice a month or more often: (a drink is one 5 ounce glass of wine or equivalent) a. ingestion of 5 drinks or more in a 2 hour period b. ingestion of 7 drinks or more in a 24 hour period
* At screening visit, CURRENTLY using any of the following interventions because of psychological distress (for example, for treatment of anxiety and/or other psychiatric condition). (These types of treatments are also prohibited during the study period.) a. participating in psychotherapy b. participating in CAM (complementary and alternative medical interventions) c. taking medication(s) (for example anxiolytics, antidepressants, and other psychotropic medications)
* Participant meets criteria for current suicidal or homicidal ideation
* Subjects who have massages on a regular basis. Regular massage usage will be defined as receiving on average 4 or more massages/year for the last 5 years
* Subjects currently employing any other CAM manual therapy and/or holistic therapies to treat a perceived health problem
* History of head injury or neurological disorder, that in the investigator's opinion would impact the data or preclude safe and successful completion of the study. - History of cancer that required chemotherapy and/or radiation treatment
* General contraindication to MRI - Because MRI uses a very strong magnet, subjects cannot have metals in their bodies or certain medical conditions. Subjects cannot have a cardiac pacemaker; hearing aid; any other implant metal in their body or eyes, including pins, screws, shrapnel, plates, teeth braces, or dentures. Subjects cannot have tattoos on their head, such as eyeliner or other permanent makeup, as they may make it impossible to get clear and usable images
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol, or complete the study
* Current participation in another research study (excluding large natural cohort trials such as 'All of Us')

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in resting state functional connectivity during fMRI | Day 1
  Resting state functional connectivity during fMRI will be evaluated immediately before and immediately after a single session of SMT or LT in healthy non-psychiatric control subjects.

SECONDARY OUTCOMES:
Change in connectivity in response to fearful/angry faces task | Day 1
  Neuronal connectivity in response to neutral/fearful/angry faces task during fMRI will be evaluated immediately before and immediately after a single session of SMT or LT in healthy non-psychiatric control subjects.
Autonomic activity (heart rate variability, heart rate, pulse) | Day 1
  Correlation of change in autonomic measures (heart rate variability, heart rate, pulse) with resting state functional connectivity and neuronal activation in response to fearful/angry faces task during fMRI will be determined immediately before and immediately after a single session of SMT or LT in healthy non-psychiatric control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rapaport, MD, Principal Investigator — Utah, University of
Locations (1):
- Huntsman Mental Health Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
We will maximize the appropriate sharing of scientific data generated from the conducted research, consistent with privacy, security, informed consent, and proprietary issues. Data management and sharing will be addressed in the informed consent process, including communicating with prospective participants how their scientific data are expected to be used and shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following peer-reviewed publication of our results, de-identified materials and data generated in the course of this project will made available upon reasonable request.
Access Criteria: Scientific data will be made accessible in a timely manner for use by the research community and the broader public. Specifically, scientific data will be made accessible as soon as possible, and no later than the time of an associated publication. We will consider relevant requirements and expectations (e.g., data repository policies, award record retention requirements, journal policies) as guidance for the minimum time frame scientific data should be made available. However, we will make scientific data available for as long as it is useful for the larger research community, institutions, and/or the broader public.